CLINICAL TRIAL: NCT02644642
Title: Utility of Disconnection Technique for One Lung Ventilation: a Comparison of a Double Lumen Endobronchial Tube With a Bronchial Blocker
Brief Title: Utility of Disconnection Technique for One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Go Un Roh, principal investigator, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AJIRB-MED-DEO-15-391
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DLT(Double Lumen Tube) group (Experimental): disconnection technique will be applied
  Interventions: Other: disconnection technique
- BB(Bronchial Blocker) group (Experimental): disconnection technique will be applied
  Interventions: Other: disconnection technique

INTERVENTIONS:
Other: disconnection technique — Before lung isolation, the ventilator stays switched-off until the carbon dioxide on the capnogram reached to zero. Then, inflate the balloon either on the double lumen tube or on the bronchial blocker.

SUMMARY:
Lung isolation technique is useful for lung or heart surgeries for better visualization. Double lumen endobronchial tube and bronchial blocker are available for lung isolation. Adding disconnection technique before lung isolation is helpful to accelerate the lung deflation. However, the utility of disconnection technique has never been evaluated in comparison of double lumen tube and bronchial blocker. Therefore, the utility of disconnection technique in two different lung isolation technique, double lumen tube and bronchial blocker will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for wedge resection for pneumothorax, unilateral
* ASA class I, II

Exclusion Criteria:

* know lung disease
* any kind of lung abnormality on preoperative chest x-ray
* coronary artery occlusive disease
* cerebrovascular disease
* pregnancy
* unable to understand the informed consent form

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Lung deflation score | 10 min after inflation of balloon
  verbal analog scale(0=no deflation, 10=complete deflation)

SECONDARY OUTCOMES:
time for initial placement | from beginning of intubation until confirmation of adequate placement with bronchoscope, approximately 5 minute
time for lung deflation | from turning the ventilator off until the carbon dioxide reach to zero on capnography, within 2 min

CONTACTS AND LOCATIONS:
Overall Officials: Go Un Roh, MD, Principal Investigator — Ajou University School of Medicine